CLINICAL TRIAL: NCT03922906
Title: Evaluation of Bowel Cleansing Using the Pure-Vu System in Patients With History of Inadequate Bowel Preparation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to COVID-19 pandemic
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL00046
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: CRC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motus Pure-Vu System (Experimental): The Pure-Vu System enables colon cleansing during standard colonoscopy using a standard colonoscope. The cleansing device, which is attached to the tip of the colonoscope and is connected to an external workstation, generates fluid jets within the colon thus dissolving the feces into small parts. The fecal matter & fluids are drained through the evacuation pipe of the cleansing device into a collecting reservoir.
  Interventions: Device: Pure-Vu System

INTERVENTIONS:
Device: Pure-Vu System — Pure-Vu System is intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating and/or cleaning the colon and evacuating the irrigation fluid (saline water), feces and other bodily fluids and matter, e.g. blood.

SUMMARY:
The study aim to evaluate the performance of Pure-Vu System in cleansing patients' colon with history of inadequate bowel preparation who are indicated for a colonoscopy procedure.

DETAILED DESCRIPTION:
The study is planned as a single arm, open trial will include up to 30 patients, aim to evaluate the performance of Pure-Vu System in cleansing patients' colon with history of inadequate bowel preparation who are indicated for a colonoscopy procedure.

Subjects will be enrolled at up to 3 clinical sites in Israel. Subjects who meet the eligibility criteria will be required to follow a standard bowel preparation instruction. Patients will be asked to record and provide their diet and bowel movements in the provided diary log at time of their scheduled colonoscopy (Diary log is provided in appendix C) and to complete a satisfaction questionnaire include feedback on the procedure and on specific aspects related to the preparation regime.

Following the procedure a telephone follow-up will be conducted at 48 hours (± 48 hours) post Pure-Vu procedure to assess patient well-being and capture any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with history of inadequate bowel preparation.
2. Subjects in the age range of 22-75 years inclusive
3. Subjects with BodyMass Index (BMI) within the range of 18.5-35 inclusive
4. Subject has signed the informed consent

Exclusion Criteria:

1. Patients with active Inflammatory Bowel Disease
2. Patients with previous history of acute diverticulitis disease or with prior incomplete colonoscopy due to diverticular disease
3. Patients with known bowel obstruction / strictures
4. History of prior surgery to colon and/or rectum
5. ASA ≥ III
6. Renal insufficiency (Creatinine ≥ 1.5mg /dL) (based on medical history)
7. Abnormal Liver enzymes (ALT/AST ≥ 2 times upper limits of normal) (based on medical history)
8. Patients taking anticoagulants drugs (excluding aspirin) or dual antiplatelet therapy
9. Patients with known coagulation disorder (INR >1.5).
10. Patients at risk of hypokalemia or hyponatremia
11. Patients with congestive cardiac failure
12. Pregnancy (as stated by patient) or breast feeding
13. Patients with altered mental status/inability to provide informed consent
14. Patients who have participated in another interventional clinical study in the last 2 months

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Boston Bowel Preparation Scale( BBPS) >1 in All Colon Segments After the Use of Pure-Vu System | Up to 2 hours
  The rating of the cleansing quality was evaluated by using the Boston Bowel Preparation Scale (BBPS), Segment score of 0-3 given to each of the 3 segments of the colon (Left side, Transverse and right side):
  Score 0- Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  Score 1- A portion of the mucosa of the colon segment is seen, but other areas of the colon segment are not seen well due to staining, residual stool, and/or opaque liquid.
  Score 2- A minor amount of residual staining, small fragments of stool, and/or opaque liquid are visible, but the mucosa of the colon segment are seen well.
  Score 3-The entire mucosa of the colon segment is seen well with no residual staining, small fragments of stool, or opaque liquid.
  subject consider as having adequate cleaning if BBPS>1 in all colon segments

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No